CLINICAL TRIAL: NCT06258694
Title: Venous Thrombo-Embolism Imaging Database
Brief Title: Venous Thrombo-Embolism Imaging Database (VTE-ID)
Acronym: VTE-ID
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC20.0326 - VTE-ID
Record Dates: First submitted 2021-01-29; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Venous Thromboembolism; Deep Vein Thrombosis; Pulmonary Embolism
Keywords: Venous thromboembolism; Image processing; Radiomics
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to identify and validate new imaging biomarkers allowing an individual phenotyping of patient with venous thrombo-embolism (VTE), mainly in terms of recurrence risk assessment and to distinguish provoked from unprovoked VTE. To do so, the investigators will create a retrospective imaging database including multiple imaging modalities, performed at diagnosis of the VTE.

DETAILED DESCRIPTION:
Using a large imaging data in VTE (including ultrasound, CT-scan and Ventilation/Perfusion lung scan), the investigators will search for association between imaging data and VTE phenotypes, mainly in terms of recurrence risk assessment and to distinguish provoked from unprovoked VTE. Then, using a radiomic approach, the investigators will try to identify new imaging biomarkers able to provide an individual phenotyping in these patients.

These imaging biomarkers will be validated using an internal cross validation technique.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Confirmed VTE diagnosis (deep vein thrombosis or pulmonary embolism).
* Inclusion in the EDITH (Etude des Déterminants et Interaction de la THrombose veineuse) between November 2009 and November 2019.
* No opposition to be included in the present study.

Exclusion Criteria:

* Patients under 18 years old.
* Patients under judicial protection.
* Patient physically or cognitively unable to give consent.
* Refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patients included in the EDITH cohort between November 2009 and Novembre 2019, with a confirmed diagnosis of VTE.
Sampling Method: Non-Probability Sample
Enrollment: 2208 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2021-02-14 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
VTE recurrence | At enrollment (retrospective follow up to 2 years)
  VTE recurrence, including Pulmonary Embolism and Deep Vein Trombosis
Distinguishing provoked from unprovoked VTE | At enrollment
  Provoked VTE is defined by the presence within the three past months, of a major risk factor (i.e. Surgery, Immobilization > 3 days, Hormonal Treatment, Pregnancy, Cancer)

SECONDARY OUTCOMES:
Individual phenotyping | At enrollment
  Correlation of the identified biomarkers with VTE phenotypes (familial history, risk factor in case of provoked VTE, and biological biomarkers as fibrinogen, D Dimeres, Hemoglobin, Platelets, CRP, heterozygous or homozygous FV Leiden, Prothrombin G20210A).

CONTACTS AND LOCATIONS:
Locations (1):
- Brest University Hospital, Brest, Finistere, France